CLINICAL TRIAL: NCT05744843
Title: Structured Exercise Versus Endovascular Reconstruction in Post Thrombotic Syndrome Pilot Study and Randomised Control Trial
Brief Title: Structured Exercise Versus Endovascular Reconstruction in Post Thrombotic Syndrome
Acronym: SEvERe-PTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 315612
Record Dates: First submitted 2023-01-25; First posted 2023-02-27 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-02

CONDITIONS: Post Thrombotic Syndrome
Keywords: deep venous; exercise; remote; stenting
MeSH Terms: conditions — Postthrombotic Syndrome; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Smartphone-based exercise arm (Experimental): Eight to twelve week smartphone delivered exercise programme
  Interventions: Behavioral: exercise
- Stenting Arm (Active Comparator): Deep venous stenting as standard of care
  Interventions: Procedure: Deep venous stenting
- Healthy Volunteers (No Intervention): Healthy Volunteers for baseline testing

INTERVENTIONS:
Behavioral: exercise — cardiovascular and lower limb strengthening exercise programme
  Other Names: remote exercise programme; smartphone-based exercise programme
  Arms: Smartphone-based exercise arm
Procedure: Deep venous stenting — Planned surgical intervention
  Other Names: Endovascular Stent reconstruction of Deep Vein
  Arms: Stenting Arm

SUMMARY:
The goal of this pilot study and randomised control trial is to compare a smartphone-based exercise programme to deep venous stenting in patients with Post Thrombotic Syndrome.

The main questions it aims to answer are:

* Is exercise as effective as stenting in these patients?
* What type of exercise is useful in these patients?
* Can exercise be used to improve the results from surgery?

Participants will be split into two groups at random. They will complete a smartphone-based exercise programme or have a deep venous stent.

They will do the following tests before and after.

* Exercise testing
* Calf muscle strength and function tests
* Ultrasound of the deep veins
* Quality of life questionnaires
* Clinical assessment of their disease

They will be compared to healthy volunteers in the pilot study. Investigators will compare exercise to stenting to see if it improves symptoms in these patients. The pilot study will help decide how many patients are needed and what exercise tests will be used for the Randomised control trial.

DETAILED DESCRIPTION:
This is a non-commercial pilot study, leading to a randomised control trial.

Primary objective:

1) To evaluate smartphone-based exercise as an alternative to stenting in patients with IVC and Iliofemoral vein outflow obstruction secondary to Post Thrombotic Syndrome (PTS).

Secondary objectives:

1. To characterise symptomatology and response to different exercise modalities in patients with chronic venous insufficiency.
2. Evaluate exercise physiology in patients with chronic venous insufficiency before and after a supervised exercise programme.
3. To explore the use of available technologies, such as smart phone applications and wearable devices to deliver a remotely monitored exercise programme.
4. To establish a method of assessment of flow (inflow and collateral flow) in patients with symptomatic venous obstruction.
5. To understand the impact of stent shape and compression on venous flow and the subsequent patient outcomes.
6. To set criteria for the stratification of patient treatment based upon objective and quantitative measures in patients with venous claudication.

Participants will be recruited to the following three groups:

Group 1. Patients with PTS that will undergo remotely supervised exercise Group 2. Patients with PTS that will undergo stenting Group 3. Healthy volunteers

All participants will undergo series of exercise tests and imaging assessments. Participants in group 1 will have these tests repeated at the end of the exercise programme, and group 2 when they attend for their six to eight week follow up visit. Participants in group 1 will be able to re-join the waiting list for stenting on the condition that they have agreement from their named consultant. Investigators anticipate all study activities to be completed before group 1 participants would have received a date for stenting, as current waiting times for stenting is in excess of 18 months.

Patients from both groups 1 and 2 will be loaned an activity tracker (FitBit) to wear. Group 1 will be asked to wear the tracker from day 1 of the exercise programme, group 2 will be asked to wear the tracker from the first post operative day. Both groups will wear the tracker until the follow up visit. This will allow measurement of general activity in both groups and allow for monitoring of compliance with exercise in group 1.

ELIGIBILITY:
Inclusion Criteria:

• Patients with symptomatic chronic venous outflow obstruction secondary to PTS or other cause affecting the Inferior Vena Cava (IVC) or iliofemoral vein(s) for greater than 12 months duration AND clinical indication for Deep Venous Stenting.

Exclusion Criteria:

* Deep Vein Thrombosis or Pulmonary Embolism within the last 12 months
* Significant or untreated left sided heart disease
* Significant or untreated respiratory disease
* Significant renal disease
* Significant liver disease
* Significant Musculoskeletal or Neurological disease
* Active cancer
* Life expectancy of less than 2 years or non-ambulatory status
* Current or Planned pregnancy within the study period
* Any other contraindication to exercise
* Any impairment preventing the provision of informed consent and compliance with study protocol
* Healthy Volunteers in the control group with presence of any arterial or venous disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Villalta score. | 1) Day 0 - baseline, prior to intervention. 2) up to 2 weeks post intervention, on average week 8-12 of the study. 3) Study completion, 6 months
  0-30, >5 diagnostic of post thrombotic disease. 5-9 is mild disease, 9-4 moderate and >15 Severe. (15 automatically added in the presence of a venous leg ulcer). Change in Villalta score

SECONDARY OUTCOMES:
VO2 max - maximal oxygen consumption | 1) Day 0 - baseline, prior to intervention. 2) up to 2 weeks post intervention, on average week 8-12 of the study.
  change in peak VO2 max on cardiopulmonary exercise testing. Increased value indicates improvement, decreased value indicates deterioration
Six minute walk test | 1) Day 0 - baseline, prior to intervention. 2) up to 2 weeks post intervention, on average week 8-12 of the study.
  change in six minute walk test. Increased distance indicates improvement, decreased distance indicates deterioration.
Incline walk test | 1) Day 0 - baseline, prior to intervention. 2) up to 2 weeks post intervention, on average week 8-12 of the study.
  Time to onset of symptoms and total incline and speed achieved. Longer time to onset, steeper incline achieved and faster speed acheived indicate improvement.
Calf ejection fraction | 1) Day 0 - baseline, prior to intervention. 2) up to 2 weeks post intervention, on average week 8-12 of the study.
  change in calf ejection fraction by plethysmography
Venous Insufficiency Epidemiological and Economic Study quality of life and symptoms (VEINES-QoL/Sym) - disease specific quality of life instrument for Chronic Venous Disorders of the Leg | 1) Day 0 - baseline, prior to intervention. 2) up to 2 weeks post intervention, on average week 8-12 of the study. 3) Study completion, 6 months
  Change in VEINES-QoL/Sym score - higher value indicates better outcome

OTHER OUTCOMES:
Maximal calf isometric contract strength as measured by isometric dynamometry. | 1) Day 0 - baseline, prior to intervention. 2) up to 2 weeks post intervention, on average week 8-12 of the study.
  Change in calf muscle maximal force output, greater output indicates improvement
deep venous flow velocity | 1) Day 0 - baseline, prior to intervention. 2) up to 2 weeks post intervention, on average week 8-12 of the study.
  changes in ultrasound assessed venous flow

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A Black, FRCS, Principal Investigator — St Thomas' Hospital
Locations (1):
- St. Thomas' Hospital, Guy's and St. Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flumignan RL, Nakano LC, Flumignan CD, Baptista-Silva JC. Angioplasty or stenting for deep venous thrombosis. Cochrane Database Syst Rev. 2025 Feb 19;2(2):CD011468. doi: 10.1002/14651858.CD011468.pub2. PMID 39968829